CLINICAL TRIAL: NCT02867982
Title: Influence of Soft Tissue Thickness and Insertion Depth of Platform Switched Implants on Crestal Bone Level Alteration
Brief Title: Platform Switched Implant and Bone Level Alteration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing University Health Science Center (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Principal Investigator, Jiang Xi, Dr., Beijing University Health Science Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I-AN-16-002
Record Dates: First submitted 2016-07-24; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Edentulous; Bone Resorption
Keywords: platform switching; crestal bone remodeling; soft tissue thickness; dental implant
MeSH Terms: conditions — Mouth, Edentulous; Bone Resorption | interventions — Dental Implants

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcrestal (Other): implants that are placed below the alveolar ridge
  Interventions: Procedure: Subcrestal implant placement; Drug: prophylactic antibiotics; Device: dental implant; Radiation: x-ray examination
- Paracrestal (Other): implants that are placed flush to the alveolar ridge
  Interventions: Procedure: Paracrestal implant placement; Drug: prophylactic antibiotics; Device: dental implant; Radiation: x-ray examination

INTERVENTIONS:
Procedure: Subcrestal implant placement — Dental implants placed 2 mm below the alveolar ridge
  Arms: Subcrestal
Procedure: Paracrestal implant placement — Dental implants placed flush to the alveolar ridge
  Arms: Paracrestal
Drug: prophylactic antibiotics — amoxicillin was used before and after implant surgery for prophylactic reasons
Device: dental implant — dental implants (Ankylos® system,Dentsply Implants Manufacturing GmbH, Mannheim, Germany) were surgically placed into the edentulous alveolar ridge
Radiation: x-ray examination — radiographies were taken before treatment and at different time point during the follow-up period

SUMMARY:
This is a two-year prospective randomized clinical study to to evaluate whether the gingival thickness and insertion depth of dental implants have any influence on marginal bone levels changes around platform switched implants.

DETAILED DESCRIPTION:
Patient selection: Patients at the Department of Oral Implantology, Peking University School and Hospital of stomatology, Bei Jing, China, who seek for implant restoration for two continous posterior teeth are potentially recruited. Inclusion criteria are generally healthy (ASA score I), non-smoking, periodontally healthy, and sufficient bone volume to place an implant without augmentation procedure. Patients were excluded in cases of medical and/or psychiatric contraindications, local infection, pregnancy or lactating, poor oral hygiene, tissue deficiency, or not willing to participate in this study.

Randomization: The two implant sites of each subject are randomly assigned to two different group with a predefined randomization tables. In order to reduce the chance of unfavorable splits between groups in terms of key prognostic factors,the randomization process will take into account the following variables: patient's gender, age, presence of adjacent teeth, distal extension sites and site location in the dental arch. Assignment will perform using a sealed envelope.

Surgical protocol: Before the surgical procedure, prophylactic antibiotics of 1g amoxicillin will prescribed to the patient 1 h before surgery, and continued with 2 g/day for 6 days. After crestal incision, full thickness buccal flap was raised, whereas lingual part was not elevated. Thickness of soft tissues was measured with 1.0-mm marked periodontal probe on the top of bone crest in the center of the two future implant sites. This ensured direct visibility of mucosal thickness during measurement. After measurements, full-thickness lingual flap is raised and subsequent implant osteotomy is finished, Two dental implants (Dentsply Implants Manufacturing GmbH, Mannheim, Germany) with diameter of 3.5 mm are ready to torch into the bone cavities. In one site (group 1), the platform of implants are placed at the crestal level (flush to the alveolar ridge) . In the other site (group 2), the implants are placed 1mm below the alveolar ridge. narrow healing abutment are connected to all the implants. The flap are repositioned and closed with interrupted single sutures. Implants are allowed for a un-submerged healing. 3 month after healing, the implant level impressions are taken, splinted restorations of two neighbouring posterior teeth are delivered 2 weeks later.

Radiographic and Clinical Examination: All the patients are required for recall visit at 3, 6,12 months and 2 years post surgery. A digital peri-apical radiograph was taken at the 1 year and 2year follow-up examination for bone level evaluation using a film holder to aim the x-ray beam perpendicular to the implant threads, and the implant length is used as calibration for the measurement. Using a image analysis software (ImageJ, version 1.47, NIH, Bethesda, MD, USA), the investigators are able to have an accurate assessment of the crest of bone and to analyze the bone changes over period of time. Bone loss was defined as a positive value and bone gain as a negative one. Mean values, standard deviations, and maximum and minimum values were calculated. Furthermore, periodontal parameters [bleeding on probing (BOP), probing pocket depth (PPD), modified plaque index on adjacent teeth and implants] were assessed.

ELIGIBILITY:
Inclusion Criteria:

* lose of two posterior teeth more than 3 months
* generally healthy (ASA score I)
* non-smoking
* periodontally healthy
* sufficient bone volume to place an implant without augmentation procedure

Exclusion Criteria:

* medical and/or psychiatric contraindication to dental implant restoration
* local infection
* pregnancy or lactating
* poor oral hygiene
* tissue deficiency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Changes of marginal bone levels of dental implant | 3 months, 6 months, 1 year and 2 years post intervention (implant surgery)
  Mesial and distal marginal bone level alterations at different time point compared with the base line. Marginal bone levels were measured with an image analysis software to the accuracy of 0.01 mm and the implant length is used as calibration for the measurement.

SECONDARY OUTCOMES:
Bleeding on probing(BOP) | 3 months, 6 months, 1 year and 2 years post intervention (implant surgery)
  bleeding index whiling probing the implant restorations
Probing pocket depth(PPD) | 3 months, 6 months, 1 year and 2 years post intervention (implant surgery)
  probing depth of implant supported restorations
modified plaque index(PI) | 3 months, 6 months, 1 year and 2 years post intervention (implant surgery)
  Modified plaque index to evaluate the oral hygiene conditions

CONTACTS AND LOCATIONS:
Overall Officials: Xi Jiang, DMD, Principal Investigator — Peking University school and hospital of stomotology, Department of oral implantology

IPD SHARING:
Plan to Share IPD: Yes